CLINICAL TRIAL: NCT05751265
Title: Tislelizumab Combined With Chemotherapy in the Cross-line Treatment of First-line Resistant Advanced Gastric Cancer, Single-arm, Exploratory Clinical Study
Brief Title: Tislelizumab Combined With Chemotherapy in the Cross-line Treatment of First-line Resistant Advanced Gastric Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fujian Cancer Hospital (Other Government)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GC-01
Record Dates: First submitted 2023-02-21; First posted 2023-03-02 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-02

CONDITIONS: Gastric Cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — tislelizumab; Fluorouracil; Paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Tislelizumab combined with chemotherapy (Experimental)
  Interventions: Drug: Tislelizumab; Drug: 5Fu; Drug: Paclitaxel injection

INTERVENTIONS:
Drug: Tislelizumab — Participants will receive Tislelizumab, 200mg, intravenously over 30 - 60 minutes, day 1 of every 3 weeks . Discontinuation will be considered due to toxicity, withdrawal of consent, or end of study. Every 3-week treatment period was considered to be a cycle.
Drug: 5Fu — Participants will receive 5-FU, 2.4 g/m2，bid，d1-d14，q3w
Drug: Paclitaxel injection — Participants will receive paclitaxel 135 mg/m2 ivgtt q2w or 175mg/m2 q3w

SUMMARY:
To explore the efficacy of Tislelizumab combined with chemotherapy in the treatment of advanced gastric cancer after first-line resistance

ELIGIBILITY:
Inclusion Criteria:

* Gastric adenocarcinoma confirmed by pathology (including histology or cytology) and locally advanced or metastatic (stage IV) tumor that is unresectable; There is no known HER2+.
* Age 18-75;
* ECOG score: 0-2;
* Patients who had previously failed first-line immunization combined with chemotherapy (oxaliplatin combined with capecitabine or FP);
* Adequate organ and bone marrow function, meeting the following definitions:

  1. Blood routine (no blood transfusion, no granulocyte colony stimulating factor [G-CSF], no other drug correction within 14 days before treatment);Absolute count of neutrophils (ANC) ≥1.5×109/L;Hemoglobin (HB) ≥9.0 g/dL;Platelet count (PLT) ≥80×109/L;
  2. Blood biochemistry Serum creatinine (Cr) ≤ 1.5× upper limit of normal (ULN) or creatinine clearance ≥60 mL/min;Serum albumin ≥2.8g/dL, for patients with poor nutritional status before neoadjuvant therapy, patients who met the requirements through parenteral nutrition could also be included in the group;Total bilirubin (TBIL) ≤ 1.5×ULN;Aspartate aminotransferase (AST) or alanine aminotransferase (ALT) level ≤2.5×ULN;
* Expected survival > 6 months;
* Fertile female subjects and male subjects whose partners are of childbearing age are required to use a medically approved contraceptive during the study treatment period and for at least 3 months after the last treatment;
* Patients who volunteered to participate in this study and signed informed consent.
* According to RECIST1.1 criteria, the patient had at least one target lesion with a measurable diameter (tumor lesion with long diameter ≥10mm, lymph node lesion with short diameter ≥15mm, scanning layer thickness 5mm);

Exclusion Criteria:

* Patients who received first-line immunotherapy for less than 3 months or experienced hyperprogression in first-line therapy or developed Grade 3 or above irAE during first-line therapy;
* Patients who have previously received other immunotherapy (including other investigational drugs) with less than 5 half-lives since the initial investigational drug use.
* Pregnant or lactating women;
* Participants who participated in other clinical studies and did not recover toxic reactions 28 days before enrollment;
* Have had other malignancies in the last 5 years or at the same time, except for cured basal cell carcinoma of the skin and carcinoma in situ of the cervix;
* Severe heart, liver, lung and kidney diseases; Neurological and mental diseases;
* The presence of uncontrolled or symptomatic active central nervous system (CNS) metastases, which may be characterized by the presence of clinical symptoms, cerebral edema, spinal cord compression meningitis, pia meningeal disease, and/or progressive growth.For patients with CNS metastases that are adequately treated and whose neurological symptoms return to baseline at least 2 weeks prior to randomization (residual signs or symptoms associated with CNS treatment can be enrolled.In addition, subjects must either stop corticosteroids or receive prednisone (or an equivalent dose of another corticosteroid) at least 2 weeks prior to randomization;
* Patients with hypertension (systolic blood pressure >140 mmHg, diastolic blood pressure >90 mmHg) who cannot be reduced to the normal range after antihypertensive medication;
* Patients with grade I or above coronary heart disease, arrhythmias (including prolonged QTc interval > 450 ms in men and > 470 ms in women), and cardiac insufficiency;
* Patients with abnormal coagulation function (INR>1.5, APTT>1.5 ULN);
* Patients with a history of cardiovascular and cerebrovascular diseases who are still taking thrombolytic drugs or anticoagulants orally.
* Presence of any active, known or suspected autoimmune disease.Subjects who are in a stable state and do not require systemic immunosuppressive therapy are admitted: e.g., type 1 diabetes, hypothyroidism requiring hormone replacement therapy only, and skin conditions requiring no systemic therapy (e.g., vitiligo, psoriasis, and alopecia).
* Concurrent autoimmune diseases or a history of chronic or recurrent immune diseases, including a history of immunodeficiency such as HIV-positive testing or a history of organ transplantation and allogeneic bone marrow transplantation.
* Patients with other concomitant diseases that, in the judgment of the investigator, seriously endanger the patient's safety or affect the patient's completion of the study;
* Patients with uncontrolled epilepsy, central nervous system disease or mental disorder whose clinical severity is judged by the investigator to be likely to prevent the signing of informed consent or have multiple factors affecting oral medication (such as inability to swallow, persistent uncontrollable nausea and vomiting, chronic diarrhea, and intestinal obstruction);
* Allergic to the test drug or its excipients;
* Persons deemed unsuitable for inclusion by the researcher.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | At the end of Cycle 3 (each cycle is 21 days)
  Objective Response Rate Determine the tumor shrinkage rate, tumor boundary and the adhesion of tumor

SECONDARY OUTCOMES:
Progression-free survival | up to 12 months
  The length of time from enrollment until the time of progression of disease